CLINICAL TRIAL: NCT00136422
Title: A Phase I Study of Vaccination With Lethally Irradiated, Autologous Acute Myeloblastic Leukemia Cells Engineered by Adenoviral Mediated Gene Transfer to Secrete Human Granulocyte-Macrophage Colony Stimulating Factor in Patients With Advanced Myelodysplasia or Acute Myelogenous Leukemia
Brief Title: Study of Vaccination With Autologous Acute Myeloblastic Leukemia Cells in Patients With Advanced Myelodysplasia or Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 99-249
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplasia
Keywords: AML; acute myelogenous leukemia; MDS; myelodysplasia; vaccine
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts

INTERVENTIONS:
Biological: autologous tumor cells

SUMMARY:
The purpose of this study is to test the safety of a new investigational acute myeloblastic leukemia (AML) vaccine and see what effects (good and bad) it has on patients with advanced myelodysplasia or acute myelogenous leukemia.

DETAILED DESCRIPTION:
This study will make use of leukemic myeloblasts harvested by bone marrow aspirate in patients with myelodysplasia and acute myelogenous leukemia. These harvested tumor cells will be modified by adenoviral mediated gene transfer to secrete granulocyte-macrophage colony stimulating factor (GM-CSF).

Patients will be administered vaccines at one of three dose levels (as determined by total cell yield). Vaccinations will be given weekly for three weeks, followed by every other week until the vaccine supply is exhausted or when patients are removed from the study.

The patient will receive a minimum of six vaccinations, but more will be administered if the vaccine is available.

During the course of the study, patients will be tested to see how their immune system is reacting to the vaccinations. Testing will include bloodwork evaluating the immune cells in the body at monthly intervals. Skin biopsies may also be performed to see if an immune reaction is occuring at the injection site.

During the first course of treatment, a bone marrow biopsy and aspirate may be performed monthly.

The length of time on this study depends upon the number of vaccines available and whether or not unacceptable side effects occur.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically documented myelodysplasia or acute myelogenous leukemia.
* The patients with myelodysplasia must also have: French-American-British (FAB) subtype refractory anemia with excess blasts (RAEB) or refractory anemia with excess blasts in transformation (RAEB-T), or normal or hypercellular bone marrow.
* The patients with acute myelogenous leukemia must also: not be candidates for myelosuppressive chemotherapy due to age or comorbid disease, or have relapsed acute myelogenous leukemia or be refractory to standard therapy and not likely to require cytoreductive therapy within 60 days
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Estimated life expectancy of 6 months or greater.
* Age at least 18 years.
* Greater than 4 weeks from any chemotherapy, radiotherapy, immunotherapy, or systemic glucocorticoid therapy (non-glucocorticoid hormonal therapy allowed).
* Greater than 2 months following bone marrow or peripheral blood stem cell transplantation or treatment with donor lymphocyte infusion (DLI).

Exclusion Criteria:

* Uncontrolled active infection.
* Pregnancy or nursing mothers.
* Previous participation in an adenovirus based trial.
* The patients with myelodysplasia who have either: FAB subtype refractory anemia (RA), refractory anemia with ringed sideroblasts (RARS), chronic myelomonocytic leukemia (CMML), or the presence of hypocellular bone marrow.
* Chemotherapy, radiotherapy, immunotherapy, or systemic steroid therapy within the last 4 weeks.
* Active central nervous system (CNS) disease.
* Evidence of infection with the human immunodeficiency virus.
* Active psychiatric or mental illness making informed consent or careful clinical follow-up unlikely.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2000-01; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of preparing lethally irradiated autologous myeloblastic leukemia cells engineered by adenoviral mediated gene transfer to secrete GM-CSF in patients with myelodysplastic syndromes (MDS) or AML

SECONDARY OUTCOMES:
To determine the safety and biologic activity of vaccination with lethally irradiated, autologous myeloblastic leukemia cells engineered by adenoviral mediated gene transfer to secrete GM-CSF in patients with MDS or AML

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. DeAngelo, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States